CLINICAL TRIAL: NCT04963777
Title: Effect of Prebiotic Fibre on Glycemic Control, Gut Microbiota, and Intestinal Permeability in Type 1 Diabetes
Brief Title: Prebiotics in Patients With Type 1 Diabetes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Principal Investigator, Dr. Raylene Reimer, Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: REB21-0852
Record Dates: First submitted 2021-07-12; First posted 2021-07-15 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-04

CONDITIONS: Type 1 Diabetes
Keywords: Gut microbiota; Glycemic control; Prebiotic; Oligofructose-enriched inulin; Hypoglycemia
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Prebiotics

STUDY DESIGN:
Intervention Model Description: Multi-centre placebo controlled double-blind randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The prebiotic and placebo are both white powders with similar sweet taste and dissolve in water.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Prebiotic (Experimental): Oligofructose-enriched inulin
  Interventions: Dietary Supplement: Prebiotic
- Placebo (Placebo Comparator): Maltodextrin
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prebiotic — Chicory root derived inulin-type fructan (13.2 kcal/day for ages 8-13 years; 26.4 kcal/day for ages ≥14 years)
  Arms: Prebiotic
Dietary Supplement: Placebo — Maltodextrin (isocaloric; 13.2 kcal/day for ages 8-13 years; 26.4 kcal/day for ≥14 years)
  Arms: Placebo

SUMMARY:
Evidence suggests that prebiotic fibre can correct dysbiosis, reduce intestinal permeability and improve glycemic control. The investigators hypothesize that microbial changes induced by prebiotics contribute to gut and endocrine adaptations that reduce glucose fluctuations, including less hyper- and hypoglycemia in type 1 diabetes (T1D). The primary objective is to compare the change in frequency of hypoglycemia from baseline to 6 months in n=144 individuals with T1D treated with a 6-month course of prebiotic or placebo as an adjunct to insulin. Secondary objectives will be aimed at understanding the mechanisms by which the prebiotics could affect glycemic control.

DETAILED DESCRIPTION:
The investigators hypothesize that, as an adjunct to insulin, prebiotic supplementation will reduce the frequency of hypoglycemia and improve glycemic variability that is accompanied by enhanced serum C-peptide levels, a reduction in intestinal permeability and systemic inflammation, and altered gut microbiota.

Primary Objective To compare the change in frequency of hypoglycemia from baseline to 6 months in individuals with T1D treated with a 6-month course of prebiotic or placebo as an adjunct to insulin.

Secondary Objectives

1. To determine the change in glycemic variability and glycemic control using Continuous Glucose Monitor (CGM) metrics including: percentage change in Time In-, Below-, and Above-Range (i.e. TIR, TBR, and TAR) and A1C from baseline to 6 months in those treated with prebiotic or placebo.
2. To compare the change in stimulated C-peptide and pro-insulin from baseline to 6 months.
3. To determine the change in IP from baseline to 6 months.
4. To determine the change in serum inflammatory markers (IL-6, IFN-gamma, TNF, C-reactive protein, and IL-10).
5. To examine quality of life (QOL) and fear of hypoglycemia ratings, and adverse reactions (severe hypoglycemia, diabetic ketoacidosis, side effects).
6. To examine prebiotic-induced changes in gut microbiota composition and function (shotgun sequencing) and their metabolic by-products (fecal and serum metabolomics).
7. To compare the change in frequency of hypoglycemia from baseline to 9 months to determine persistence of effects post-intervention.
8. To determine the change in glycemic variability from baseline to 9 months to determine persistence of effects post-intervention.

ELIGIBILITY:
Inclusion Criteria:

Lead Site:

* Diagnosed with type 1 diabetes (based on Diabetes Canada 2018 Clinical Practice Guideline diagnostic criteria) in the previous 12 months.
* Age 7 years and above (as per our pilot trial and able to complete the required tests).

Subsites:

* Diagnosed with type 1 diabetes (based on Diabetes Canada 2018 Clinical Practice Guideline diagnostic criteria) in the previous 12 months.
* Age 7 to 17 years of age.

Exclusion Criteria:

* Regular use of medications or supplements that could affect gut microbiota (examples: antibiotics, probiotic or prebiotic supplements, laxatives) within 3 months prior to enrollment.
* Previous intestinal surgery.
* Another chronic medical condition that could affect gut microbiota or intestinal permeability (examples: Crohn's disease, Celiac disease, colitis, irritable bowel syndrome)
* Presence of active infection, pregnancy or lactation.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2022-03-29 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change in frequency of hypoglycemia | 6 months
  Blood glucose <3.9 mmol/L from continuous glucose monitor data

SECONDARY OUTCOMES:
Change in glycemic variability | 6 months
  CGM-recorded composite of percentage of 'time-in-range" (glucose of 3.9-10 mmol/L), "time-below-range" as mild (glucose 3.0-3.9 mmol/L) or moderate (glucose <3.0 mmol/L) hypoglycemia, and "time-above- range" as moderate (glucose 10.1-13.9 mmol/L) and severe (glucose >13.9 mmol/L) hyperglycemia.
Change in glycemic control | 6 months
  Glycated hemoglobin (A1C)
Change in stimulated C-peptide | 6 months
  Serum collected during a mixed meal tolerance test
Change in serum proinsulin | 6 months
  Serum collected during a mixed meal tolerance test
Change in Intestinal permeability | 6 months
  Urinary lactulose/mannitol test
Change in lipopolysaccharide | 6 months
  Serum lipopolysaccharide concentration
Change in Inflammatory marker IL-6 | 6 months
  Serum IL-6
Change in Inflammatory marker IFN-γ | 6 months
  Serum IFN-γ
Change in Inflammatory marker TNF | 6 months
  Serum TNF
Change in Inflammatory marker CRP | 6 months
  Serum CRP
Change in Inflammatory marker IL-10 | 6 months
  Serum IL-10
Change in quality of life | 6 months
  Diabetes-specific quality of life survey
Change in fear of hypoglycemia | 6 months
  Fear of hypoglycemia ratings survey
Change in gut microbiota composition | 6 months
  Fecal microbiota taxonomy
Change in gut microbiota function | 6 months
  Fecal microbiota shotgun sequencing
Change in serum metabolite concentration | 6 months
  Serum LC-Qtof-Mass Spec metabolomics
Change in fecal metabolite concentrations | 6 months
  Serum LC-Qtof-Mass Spec metabolomics
Change in frequency of hypoglycemia post-intervention | 9 months
  Blood glucose <3.9 mmol/L from continuous glucose monitor data
Change in glycemic variability post-intervention | 9 months
  CGM-recorded composite of percentage of 'time-in-range" (glucose of 3.9-10 mmol/L), "time-below-range" as mild (glucose 3.0-3.9 mmol/L) or moderate (glucose <3.0 mmol/L) hypoglycemia, and "time-above- range" as moderate (glucose 10.1-13.9 mmol/L) and severe (glucose >13.9 mmol/L) hyperglycemia.
Change in glycemic control post-intervention | 9 months
  Glycated hemoglobin (A1C)

OTHER OUTCOMES:
Change in dietary intake | 6 months
  24 hour dietary recall (energy intake, kcal)
Change in dietary intake | 6 months
  24 hour dietary recall (fat intake, grams)
Change in dietary intake | 6 months
  24 hour dietary recall (carbohydrate intake, grams)
Change in dietary intake | 6 months
  24 hour dietary recall (protein intake, grams)
Change in dietary intake | 6 months
  24 hour dietary recall (fiber intake, grams)

CONTACTS AND LOCATIONS:
Overall Officials: Raylene A Reimer, PhD, RD, Principal Investigator — University of Calgary
Locations (3):
- Canada (3):
  - University of Calgary, Calgary, Alberta
  - University of Alberta, Edmonton, Alberta
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No
De-identified participant data will be available from the corresponding author upon reasonable request.

REFERENCES:
- [Derived] Huang C, Rosolowsky E, Nour MA, Butalia S, Ho J, Mayengbam S, Wang W, Pyke S, Virtanen H, Reimer RA. Prebiotic supplementation in patients with type 1 diabetes: study protocol for a randomised controlled trial in Canada. BMJ Open. 2025 May 31;15(5):e102486. doi: 10.1136/bmjopen-2025-102486. PMID 40449951